CLINICAL TRIAL: NCT04007809
Title: Phenotypic and Genotypic Characterization of a Cohort of Pediatric Patients With New-onset Type 1 Diabetes
Brief Title: Phenotypic and Genotypic Characterization of New-onset Type I Diabetes
Acronym: DIATAG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Fonds National de la Recherche Scientifique (Other); BESPEED (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DIATAG
Record Dates: First submitted 2019-06-03; First posted 2019-07-05 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Type1diabetes
Keywords: type 1 diabetes; children; biomarkers
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Glucagon; Glucagon-Like Peptide 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- New-onset Type 1 diabetes (Experimental)
  Interventions: Other: Glucagon

INTERVENTIONS:
Other: Glucagon — Every patients will undergo stimulated C peptide test. Glucagon will be administered using intravenous route (0,03 mg/kg, max 1mg).
  Other Names: Glucagen

SUMMARY:
The goal of DIATAG study is the identification of biomarkers of T1D evolution in a pediatric cohort.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is a common chronic disease in childhood. Clinical presentation at onset of T1D can vary among patients from long-standing diabetes triad symptoms (polyuria, polydipsia and weight loss) to coma and ketoacidosis. The initial clinical presentation of T1D was shown to have long-term influence on glycemic control of the patient. The investigators initiated a collaborative consortium including six pediatric clinics in Belgium to better characterize new-onset T1D patients.

Hypothesis :

1. Different subgroups of T1D patients might exist, underlying different physiopathology of T1D :

   * The investigators will first investigate the presence of biomarkers in different fluids (e.g. urine, blood, feces,...).
   * The investigators will correlate results with clinical parameters of glycemic control. Dynamic tests (HOMA and stimulated C peptide) will be realized at 2 defined time points of the follow-up.
2. Glucose variability can be influenced by external factors (e.g. diet, physical activity, Quality of Life (QoL),...) The investigators will evaluate those external factors using approved questionnaires. They will presented to the patient and its parents at 2 defined time points.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes de novo according to American Diabetes Association criteria:

   1. Polyuria, polydipsia, weight loss ± ketoacidosis
   2. Fasting blood glucose ≥126 mg/dL AND/OR blood glucose ≥200 mg/dL at the 120th minute of an Oral Glucose Tolerance Test (OGTT) AND/OR HbA1c ≥6.5% AND/OR a patient with symptoms of hyperglycemia/hyperglycemic crisis (see 8. a. 2.) with random blood glucose ≥200 mg/dL.
   3. Presence in the serum of one or more anti-islet autoantibodies (anti-insulin, anti-IA2, anti-GAD65, anti-ZnT8)
2. Age between 6 months and 18 years.
3. Male or female.
4. Positive for one or more autoantibodies typically associated with Type 1 Diabetes (TD1).
5. Free written and oral consent.

Exclusion Criteria:

1. Children under 6 months of age.
2. Treatment that interferes with insulin secretion and insulin sensitivity (e. g. sulfonylureas, diazoxide, somatostatin, methylxanthine derivatives, corticosteroids, biguanide, incretins).
3. Presence of celiac disease (diagnosis based on pathological duodenal biopsy), recently diagnosed (within 1 month), at the time of inclusion.
4. Autoimmune/auto-inflammatory disease (other than type 1 diabetes) or active malignant disease present at inclusion.
5. Obesity defined by a Body Mass Index (BMI) with a z-score >+3 Standard Deviation.
6. Hepatic, renal or adrenal insufficiency.
7. History of spinal cord allograft.
8. History of post-hemolytic-uremic diabetes.
9. Absence of anti-pancreatic islet auto-antibodies.
10. Dysmorphic with suspicion of underlying genetic syndrome.
11. Participation in another study within the previous 3 months, with administration of blood derivatives or potentially immunomodulating treatments.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of T1D subgroups by using follow-up of clinical parameters : weight in kilograms | up to 18 months after diagnosis
  weight in kilograms
Evaluation of T1D subgroups by using follow-up of clinical parameters : Height in centimeter | up to 18 months after diagnosis
  Height in centimeter
Evaluation of T1D subgroups by using follow-up of clinical parameters : Body mass index (kg/m²) | up to 18 months after diagnosis
  Body mass index (kg/m²)
Evaluation of T1D subgroups by using follow-up of clinical parameters : glycemic variability (%) | up to 18 months after diagnosis
  glycemic variability (%)
Follow-up of laboratory results - glycemia (mg/dL) | up to 18 months after diagnosis
  glycemia (mg/dL)
Follow-up of laboratory results - Insulin (mUI/L) | up to 18 months after diagnosis
  Insulin (mUI/L)
Follow-up of laboratory results - HbA1C (%) | up to 18 months after diagnosis
  HbA1C (%)
Follow-up of laboratory results - C-peptide (mUI/L) | up to 18 months after diagnosis
  C-peptide (mUI/L)
Evaluation and follow-up of diet, physical activity, quality of life using validated questionnaires. | up to 18 months after diagnosis
  Composite of Physical Activity Questionnaire (PAQ), DisabKids, Health Behaviour in School-aged Children (HBSC)
Evaluation and follow-up of physical activity | up to 18 months after diagnosis
  Physical Activity Questionnaire (PAQ). This questionnaire consists of 8 items. Once you have a value from 1 to 5 for each of the 8 items (items 1 to 8) used in the Physical Activity composite score, you simply take the mean of these 8 items, which results in the final PAQ activity summary score.
  A score of 1 indicates low physical activity, wheareas a score of 5 indicates high physical activity.
Evaluation and follow-up of quality of life: DisabKids Questionnaires | up to 18 months after diagnosis
  DisabKids Questionnaires. The paper version of DISABKIDS consisted of the generic health related quality of life questionnaire for 8- to 18-year-olds (37 items) and the DISABKIDS Diabetes module (10 items). The questionnaire is designed to measure health related quality of life of children with a chronic medical condition. Questions are answered on a Likert type scale of 1-5 points. Lower scores correspond to better quality of life.

SECONDARY OUTCOMES:
Production of prediction model of β-cell mass evolution | up to 18 months after diagnosis
  Composite score using clinical parameters and laboratory results

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Polle OG, Delfosse A, Martin M, Louis J, Gies I, den Brinker M, Seret N, Lebrethon MC, Mouraux T, Gatto L, Lysy PA; DIATAG Working Group. Glycemic Variability Patterns Strongly Correlate With Partial Remission Status in Children With Newly Diagnosed Type 1 Diabetes. Diabetes Care. 2022 Oct 1;45(10):2360-2368. doi: 10.2337/dc21-2543. PMID 35994729